CLINICAL TRIAL: NCT02450474
Title: Pilot Evaluation of Intermittent Pneumatic Compression and Neuromuscular Electrical Stimulation for Enhancing Vascular Refilling in Haemodialysis
Brief Title: Mobilising Lower Limb Fluid for Hemodynamic Stability in Haemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RL14/11224
Record Dates: First submitted 2014-12-16; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: baseline - IPC (Other): A: baseline - IPC - washout - NMES - washout - follow up
  The baseline phase, washout phase and follow up phase will consist of treatment as normal. IPC phase will consist of normal care plus IPC of the lower limbs for the duration of each dialysis session.
  Interventions: Device: Intermittent pneumatic compression device; Device: Neuromuscular electrical stimulation
- B: baseline - NMES (Other): B: baseline - NMES - washout - IPC - washout follow up
  The baseline phase, washout phase and follow up phase will consist of treatment as normal. NMES phase will consist of normal care plus stimulation of the foot and calf muscles for a period of one hour during dialysis.
  Interventions: Device: Intermittent pneumatic compression device; Device: Neuromuscular electrical stimulation

INTERVENTIONS:
Device: Intermittent pneumatic compression device — Flowtron, Circulation Booster and Sports XL devices will be used.
Device: Neuromuscular electrical stimulation — Flowtron, Circulation Booster and Sports XL devices will be used.

SUMMARY:
Cardiovascular disease is the leading cause of death of dialysis patients and poor fluid management is associated with the increased risk. One of the principal limitations in avoiding chronic fluid overload in this patient group is the refilling rate the rate at which fluid is transferred from tissues into the vascular system. If this rate cannot match the prescribed rate of fluid removal during dialysis the patient will end up with chronic fluid overload.

Two proposed methods of increasing the rate of refilling are intermittent pneumatic compression (IPC) devices, which increase the pressure of the fluid in tissue, and neuromuscular electrical stimulation (NMES) which activates the muscle pump and lymphatic drainage.

This investigation will trial the use of these two methods in patients suspected of having inadequate refilling rates. Outcome measures will be based on fluid status, presence of oedema and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Presence of lower limb oedema as defined by pitting
* Average post dialysis fluid overload in relation to target weight greater than 0.5 litres
* Greater than one dialysis session that included an intradialytic hypotensive episode in the previous month, defined by saline influsion or nursing intervention

Exclusion Criteria:

* Less than 18 years of age
* Less than 3 months dialysis vintage
* Presence of metal implants, amputations or the inability to be weighed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Fluid Status (Body composition monitor measurement of fluid status) | Weekly
  Body composition monitor measurement of fluid statu
Quality of Life (Validated Kidney Disease Quality of Life (KDQOL36) quality of life measurement questionnaire and patient symptom questionnaire) | Weekly
  Validated KDQOL36 quality of life measurement questionnaire and patient symptom questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom